CLINICAL TRIAL: NCT01024569
Title: Mental Illness Self-Management Through Wellness Recovery Action Planning In Ohio
Brief Title: Randomized Controlled Trial of Wellness Recovery Action Planning
Acronym: WRAP RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency); Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Judith A. Cook, Professor of Psychiatry, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2006-0103; UIC WRAP Study (Other Grant/Funding Number: H133B050003)
Record Dates: First submitted 2009-12-02; First posted 2009-12-03 (Estimated); Results first posted 2020-01-10 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-12

CONDITIONS: Mental Disorders
Keywords: Severe Mental Illness; Recovery; Psychiatric Disability; Wellness; Peer Service; WRAP
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wellness Recovery Action Planning (WRAP) (Experimental): WRAP consists of 8 sessions lasting for 2-½ hours, convened once a week over a period of 8 weeks. Topics include: Introduction to WRAP, Developing a Wellness Toolbox, Creating a Daily Maintenance Plan, Identifying Triggers, Identifying Early Warning Signs, Managing When Things Break Down, and Crisis Planning. Coursework is interactive, using lecture, question and answer, group discussion, and individual or group exercises. Each session includes a lecture on recovery topics such as self-esteem, changing negative thoughts to positive ones, peer support, and lifestyle issues.
  Interventions: Behavioral: Wellness Recovery Action Planning (WRAP)
- Comparison Wait-List Group (No Intervention): Participants assigned to the comparison group were in a delayed treatment condition in which they continued in public services as usual, but were offered the chance to attend WRAP groups after their final research interview.

INTERVENTIONS:
Behavioral: Wellness Recovery Action Planning (WRAP) — WRAP consists of 8 sessions lasting for 2-½ hours, convened once a week over a period of 8 weeks.
  Arms: Wellness Recovery Action Planning (WRAP)

SUMMARY:
The purpose of this research study is to test the effectiveness of a standardized peer-led intervention to teach self-management skills in improving outcomes of individuals with a severe mental illness. The intervention is known as Wellness Recovery Action Planning or WRAP, co-developed by Dr. Mary Ellen Copeland. The focus of the inquiry is on whether and how developing an individualized plan for successful living: 1) lowers psychiatric symptoms; 2) enhances psychosocial outcomes such as self-perceived recovery, empowerment, self-advocacy, coping, and social support; 3) increases knowledge of personal mental illness self-management strategies; and 4) enhances satisfaction with the service delivery system. The study evaluated the following hypotheses:

Hypothesis #1: Compared to wait-list control subjects, those who participate in the WRAP intervention will report reduced levels of psychiatric symptoms.

Hypothesis #2: Compared to wait-list control subjects, those who participate in the WRAP intervention will report enhanced enhanced feelings of empowerment, hope, recovery, quality of life, and functioning.

Hypothesis #3: Compared to wait-list controls, those who participate in the WRAP intervention will report increased levels of social support.

Hypothesis #4: Compared to wait-list controls, those who participate in the WRAP intervention will report increased use of peer services, higher satisfaction with services, and have lower overall service costs.

Hypothesis #5: Compared to controls, those who participate in the WRAP intervention will report increased knowledge of mental illness self-management, including making/using a WRAP plan.

Hypothesis #6: There will be no difference in employment rates of control vs. intervention subjects.

DETAILED DESCRIPTION:
Eligibility criteria included having a diagnosis of serious mental illness and experiencing severe functional impairment in one or more life roles. All study participants completed telephone interviews at three points in time: study entry (pre-intervention); 8-weeks later (immediate post-intervention); and 6-months after intervention (approximately 8 months after study entry). Blinded interviewers administered valid and reliable outcome assessments that measured changes in subjects' knowledge about mental illness; emotional well-being; empowerment; hopefulness; quality of life, and functioning. All study participants were compensated for their time at each interview. All WRAP facilitators were people in recovery from serious mental illnesses who were certified and experienced WRAP facilitators. Fidelity to the WRAP curriculum was assessed on an ongoing basis throughout the study.

ELIGIBILITY:
Inclusion Criteria

* age 18 years or older
* English speaking
* severe mental illness as confirmed by: 1) a Kessler Self-Report Measure (K-6) score of 13 or higher; and/or 2) enrolled as a client of the public mental health system in the state of Ohio.

Exclusion Criteria

* non English speaking
* not meeting clinical criteria for severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2007-12; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith A. Cook, PhD, Principal Investigator — University of Illinois at Chicago, Department of Psychiatry
Locations (1):
- University of Illinois at Chicago, Department of Psychiatry, Chicago, Illinois, United States

REFERENCES:
- [Result] Cook JA, Copeland ME, Jonikas JA, Hamilton MM, Razzano LA, Grey DD, Floyd CB, Hudson WB, Macfarlane RT, Carter TM, Boyd S. Results of a randomized controlled trial of mental illness self-management using Wellness Recovery Action Planning. Schizophr Bull. 2012 Jun;38(4):881-91. doi: 10.1093/schbul/sbr012. Epub 2011 Mar 14. PMID 21402724
- [Result] Cook JA, Copeland ME, Floyd CB, Jonikas JA, Hamilton MM, Razzano L, Carter TM, Hudson WB, Grey DD, Boyd S. A randomized controlled trial of effects of Wellness Recovery Action Planning on depression, anxiety, and recovery. Psychiatr Serv. 2012 Jun;63(6):541-7. doi: 10.1176/appi.ps.201100125. PMID 22508435
- [Result] Jonikas JA, Grey DD, Copeland ME, Razzano LA, Hamilton MM, Floyd CB, Hudson WB, Cook JA. Improving propensity for patient self-advocacy through wellness recovery action planning: results of a randomized controlled trial. Community Ment Health J. 2013 Jun;49(3):260-9. doi: 10.1007/s10597-011-9475-9. Epub 2011 Dec 14. PMID 22167660
- [Result] Snyder CR, Sympson SC, Ybasco FC, Borders TF, Babyak MA, Higgins RL. Development and validation of the State Hope Scale. J Pers Soc Psychol. 1996 Feb;70(2):321-35. doi: 10.1037//0022-3514.70.2.321. PMID 8636885
- [Result] Scanlan JN, Hancock N, Honey A. The Recovery Assessment Scale - Domains and Stages (RAS-DS): Sensitivity to change over time and convergent validity with level of unmet need. Psychiatry Res. 2018 Mar;261:560-564. doi: 10.1016/j.psychres.2018.01.042. PMID 29407723
- [Result] Brashers DE, Haas SM, Neidig JL. The patient self-advocacy scale: measuring patient involvement in health care decision-making interactions. Health Commun. 1999;11(2):97-121. doi: 10.1207/s15327027hc1102_1. PMID 16370972
- [Result] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- See also: University of Illinois at Chicago National Research & Training Center — http://www.cmhsrp.uic.edu/nrtc/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wellness Recovery Action Planning (WRAP) | Comparison Wait-List Group
Started | 276 | 279
Completed | 251 | 268
Not Completed | 25 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wellness Recovery Action Planning (WRAP) | Comparison Wait-List Group | Total
Number analyzed (Participants) | 251 | 268 | 519
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (9.8) | 45.8 (9.9) | 45.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 168 | 174 | 342
  Male | 83 | 94 | 177
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 9 | 15
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 76 | 70 | 146
  White | 167 | 186 | 353
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 251 | 268 | 519
Study Site [Count of Participants; unit: Participants]
  Canton | 38 | 43 | 81
  Cleveland | 51 | 47 | 98
  Columbus | 52 | 55 | 107
  Dayton | 12 | 14 | 26
  Lorain | 53 | 57 | 110
  Toledo | 45 | 52 | 97
Diagnostic and Statistical Manual Diploma in Social Medicine (DSM-IV) Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia | 29 | 29 | 58
  Schizoaffective | 26 | 21 | 47
  Bipolar | 95 | 93 | 188
  Depressive | 60 | 65 | 125
  Other | 34 | 42 | 76
  Missing | 7 | 18 | 25

OUTCOME MEASURES:

1. Primary Outcome: Psychiatric Symptoms Recovery Using the Brief Symptoms Inventory (BSI)
Description: The BSI is a patient self-report mental health symptoms research instrument (Piersma et al., 1994). Respondents are asked how much they were bothered in the past week by 53 symptoms on 9 dimensions with a 5-point response scale ranging from ''not at all'' to ''extremely.'' We assessed the BSI Positive Symptom Score which captures the number of symptoms endorsed in a pathological direction, representing the total volume of different symptoms reported to be present to any degree. The minimum value is 0 and the maximum score is 212, where higher scores mean a worse outcome.
Time Frame: Study entry (pre-intervention), 8-weeks later (post-intervention), & 6-months after intervention (approx. 8 months after study entry)
Measure: Mean (Standard Deviation); unit: symptom severity score
Groups:
- Experimental: Received intervention
- Control: Did not receive intervention
Arm/Group | Experimental | Control
Number analyzed (Participants) | 251 | 268
symptom severity score
  Baseline | 20.6 (14.67) | 19.29 (14.09)
  Postintervention 1 | 19.52 (13.74) | 21.38 (13.68)
  Postintervention 2 | 12.20 (15.22) | 12.65 (15.00)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.027, Mixed Effects Random Regression; MIXREG Estimate = -1.16, Standard Error of Mean -2.21

2. Primary Outcome: Hopefulness
Description: Hopefulness is measured by the State Hope Scale. Hopefulness as a cross-situational long-term trait is assessed via patient self-report using a 12-item scale assessed on a 4-point Likert response scale with options ranging from "definitely false" to "definitely true" and summed to produce a total score and sub-scale scores. The minimum value for this scale is 12 and the maximum value is 48. Higher scores indicate a better income.
Time Frame: as for outcome 1
Population: The Overall Number of Participants Analyzed reflects the number of participants at Time 1/Baseline.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Wellness Recovery Action Planning (WRAP) | Comparison Wait-List Group
Number analyzed (Participants) | 248 | 264
Score on a Scale
  Baseline | 21.67 (4.66) | 21.87 (4.42)
  Post-intervention 1: number analyzed (Participants) | 221 | 228
  Post-intervention 1 | 22.47 (4.39) | 22.07 (4.06)
  Post-intervention 2: number analyzed (Participants) | 212 | 222
  Post-intervention 2 | 22.76 (4.68) | 22.16 (4.21)
Statistical Analysis 1: Comparison: Wellness Recovery Action Planning (WRAP) vs Comparison Wait-List Group; Mixed Effects Random Regression analysis was used to assess the effects of study condition on Hope outcomes; Test type: Superiority; p = 0.020, Mixed Effects Random Regression; MIXREG Estimate = 0.40, Standard Error of Mean 2.37

3. Primary Outcome: Patient Self-Advocacy
Description: The ability to advocate for oneself with medical care providers is assessed via self-report using The Patient Self-Advocacy Scale, an 18-item scale with a 5-point Likert response set ranging from "strongly disagree" to "strongly agree". Dimensions include in patient knowledge, assertiveness, and potential for mindful non-adherence to treatment. Values range from a minimum of 18 to a maximum of 90, with higher scores indicating a better outcome.
Time Frame: as for outcome 1
Population: The Overall Number of Participants Analyzed reflects the number of participants at Time 1/Baseline
Measure: Mean (Standard Error); unit: Score on a Scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 251 | 268
Score on a Scale
  Baseline (Time 1) | 3.47 (0.50) | 3.46 (0.53)
  Post-intervention 1 (Time 2): number analyzed (Participants) | 224 | 234
  Post-intervention 1 (Time 2) | 3.61 (0.52) | 3.53 (0.53)
  Post-intervention 2 (Time 3): number analyzed (Participants) | 220 | 227
  Post-intervention 2 (Time 3) | 3.65 (0.52) | 3.55 (0.49)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.029, Mixed Effects Random Regression; MIXREG Estimate = 0.05, Standard Error of Mean 0.02

4. Primary Outcome: Recovery From Mental Illness
Description: This outcome is measured by the Recovery Assessment Scale (RAS). Recovery is a psychosocial outcome assessed via patient self-ratings on a 41-item scale using a 5-point Likert-Response format ranging from "strongly disagree" to "strongly agree". The minimum value for the RAS is 41 and the maximum is 205, with higher scores indicating a better outcome. Dimensions of recovery include personal confidence and hope, willingness to ask for help, goal and success orientation, reliance on others, and not being dominated by one's residual psychiatric symptoms.
Time Frame: as for outcome 1
Population: The Overall Number of Participants Analyzed reflects the number of participants at Time 1/Baseline.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 248 | 265
score on a scale
  Baseline (Time 1) | 88.2 (14.9) | 87.4 (13.2)
  Post-intervention 1 (Time 2): number analyzed (Participants) | 222 | 231
  Post-intervention 1 (Time 2) | 92.9 (14.2) | 90.0 (13.7)
  Post-intervention 2 (Time 3): number analyzed (Participants) | 217 | 222
  Post-intervention 2 (Time 3) | 93.7 (14.7) | 91.2 (13.1)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.042, Mixed Effects Random Regression; MIXREG Estimate = 1.06, Standard Error of Mean 0.52

5. Secondary Outcome: Quality of Life Brief Assessment
Description: Quality of Life was assessed by the World Health Organization Quality of Life Brief Assessment (WHOQOL-BREF). The 8-item environment sub-scale was utilized for our study. Respondents rate their experience of 8 quality indicators over the past 2 weeks using a 5-point Likert response scale. The minimum value is 8 and the maximum is 40, with higher scores meaning better outcomes.
Time Frame: as for outcome 1
Population: The Overall Number of Participants Analyzed reflects the number of participants at Time 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Experimental | Control
Number analyzed (Participants) | 251 | 268
Score on a Scale
  Baseline (Time 1) | 13.1 (2.94) | 13.1 (2.74)
  Post-intervention 1 (Time 2): number analyzed (Participants) | 224 | 234
  Post-intervention 1 (Time 2) | 13.7 (2.97) | 13.5 (2.79)
  Post-intervention 2 (Time 3): number analyzed (Participants) | 212 | 219
  Post-intervention 2 (Time 3) | 14.1 (2.83) | 13.4 (2.97)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = .001, Mixed Effects Random Regression; MIXREG Estimate = 0.39, Standard Error of Mean 0.11

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Wellness Recovery Action Planning (WRAP) | Comparison Wait-List Group
All-Cause Mortality (participants affected / at risk) | 4/268 | 6/251
Serious Adverse Events (participants affected / at risk) | 0/268 | 0/251
Other Adverse Events (participants affected / at risk) | 1/268 | 1/251
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wellness Recovery Action Planning (WRAP) (N=268) | Comparison Wait-List Group (N=251)
Psychiatric Disorders (Psychiatric disorders) | 1 (1) | 0 (0) — At the Time 2 interview, subject mentioned that she had been thinking about harming herself and had been feeling this way for several weeks. The interviewer activated the study's crisis protocol and followed up with subject.
Psychiatric Disorders (Psychiatric disorders) | 0 (0) | 1 (1) — At the Time 1 interview, subject responded that she had been "a little bothered" by suicidal thoughts during the past week, due to the recent death of her daughter. The study's crisis protocol was activated and subject was followed up with.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes